CLINICAL TRIAL: NCT07398027
Title: Post-Market Study of Transbronchial Cryo-assisted RFA During Robotic Assisted Bronchoscopy With Subsequent Surgical Resection (CRONOS-CH)
Brief Title: Post-Market Study of Transbronchial Cryo-assisted RFA During Robotic Bronchoscopy With Subsequent Surgical Resection
Acronym: CRONOS-CH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carolin Steinack (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor-Investigator, Carolin Steinack, Head of Interventional Pulmonology, Sponsor, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 639001022
Record Dates: First submitted 2026-01-21; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm clinical investigation conducted at a single site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HybridTherm Cryo-Assisted RFA & surgical resection (Experimental): Participants undergo transbronchial cryo-assisted radiofrequency ablation (RFA) using the CE-marked HybridTherm® system during routine diagnostic bronchoscopy. When clinically indicated, mediastinal lymph node staging by performed. Surgical resection of the treated lung lesion follows according to the standard clinical treatment plan.
  Interventions: Device: HybridTherm® System

INTERVENTIONS:
Device: HybridTherm® System — Transbronchial cryo-assisted radiofrequency ablation (RFA) performed using the CE-marked HybridTherm® system during routine diagnostic bronchoscopy, within the intended use of the device.

SUMMARY:
The purpose of this study is to confirm the procedural feasibility and device usability of the HybridTherm® system during bronchoscopic cryo-assisted radiofrequency ablation (RFA) performed prior to scheduled surgical resection in patients with lung cancer. The bronchoscopy session includes tumor ablation and, when clinically indicated, mediastinal lymph node staging by EBUS-TBNA.

DETAILED DESCRIPTION:
This is a prospective, single-arm, post-market clinical investigation conducted in Switzerland to collect clinical data on the use, safety, and performance of the CE-marked HybridTherm® system during routine bronchoscopic tumor management procedures. The investigation is classified as a ClinO-MD Category A1 medical device study, as the HybridTherm® system is CE-marked and used strictly within its intended purpose under normal conditions of clinical use.

The investigation is investigator-initiated and single-center, conducted at the University Hospital Zurich. The Sponsor-Investigator is responsible for the initiation, conduct, management, safety oversight, and data handling of the study in accordance with the Swiss Human Research Act (HRA), the Ordinance on Clinical Trials with Medical Devices (ClinO-MD), ISO 14155, and applicable ethical requirements. Ethics Committee approval is required prior to study initiation, and the investigation will begin only after a positive written decision from the competent cantonal ethics committee has been obtained.

The HybridTherm® system is a bipolar cryo-cooled radiofrequency ablation device intended for incision, coagulation, and ablation of tissue during flexible endoscopic procedures in the tracheobronchial system. The system provides internally cooled radiofrequency energy to delay tissue desiccation and impedance rise, thereby enabling controlled energy delivery during ablation. In this investigation, the device is used during clinically indicated bronchoscopic procedures without deviation from its approved indication or standard clinical workflow.

All enrolled participants undergo diagnostic bronchoscopy as part of routine clinical care, including mediastinal lymph node staging when clinically indicated. Transbronchial cryo-assisted radiofrequency ablation is performed during the same bronchoscopy session under general anesthesia. Surgical resection of the targeted lung lesion follows according to the established oncologic treatment plan and is not altered by study participation. No randomization, blinding, or comparator intervention is included.

Data collected in this investigation are derived exclusively from standard-of-care procedures, routine imaging, device readouts, and histopathological assessment of resected specimens. No additional diagnostic tests, therapeutic interventions, or protocol-mandated procedures beyond routine clinical practice are introduced. All analyses are descriptive in nature and are intended to support post-market evaluation of procedural feasibility, safety, and device usability.

The investigation is designed to generate clinical experience and safety data that may inform future clinical research and support the continued evaluation of bronchoscopic cryo-assisted radiofrequency ablation using the HybridTherm® system within standard treatment pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require diagnostic bronchoscopy for suspicious lung lesions with mediastinal lymph node status confirmed as NO by one of the following: Prior PET-CT showing no FDG-avid mediastinal lymph nodes, OR intraoperative EBUS-TBNA with ROSE confirming negative lymph nodes (performed when clinically indicated per section 6.1).
* Solitary pulmonary lesions ≤ 2.5cm with histologically or cytologically confirmed primary lung cancer.
* Suitable candidate for surgical resection of the tumor targeted for ablation
* Interdisciplinary tumor board consent
* Ability to read, understand, and sign patient Informed Consent Form (ICF)
* Age ≥ 18-years-old
* ≥ 20 mm of free space between the calculated intended ablation zone and the lung parenchyma or any critical structures (pleura, vessels and main bronchi).

Exclusion Criteria:

* Pregnant or nursing (breast feeding) females
* Central tumors abutting vital structures (main bronchus, pulmonary artery, esophagus, trachea)
* Thoracic electronic implants (e.g., pacemakers, ICDs)
* Uncorrectable coagulopathy or platelet count ≤ 50,000/mm³
* Patients receiving anticoagulant therapy or with pulmonary hypertension that, in the opinion of the Investigator, poses an unacceptable safety risk for bronchoscopy and ablation.
* Severe, uncontrolled comorbidities
* Active systemic infection
* Prior radiation therapy (SBRT) in the intended ablation zone
* Recent Investigational therapy within the last 30 days that the investigator deems could interfere with proceeding in the clinical investigation
* Tumors associated with atelectasis, obstructive pneumonitis, pleural effusion, or fibrosis
* Investigators determine that study participation poses safety risk
* Any comorbidities judged by the principal Investigator to be contraindicated for bronchoscopy
* Subject was judged unsuitable for study participation by the Investigator for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successful Completion of Bronchoscopic Cryo-assisted RFA Using the HybridTherm® System | Day 0 (Diagnostic Bronchoscopy and RFA Procedure)
  Successful device use, defined as the completion of ablation with the HybridTherm® system with investigator confirmation that the ablation zone achieved sufficient coverage based on intra-procedural imaging
Number of Participants with Bleeding-Related Serious Adverse Events Associated with the Investigational Device and/or RFA Procedure | From Day 0 (Diagnostic Bronchoscopy and RFA Procedure) through End of Study (6-7 weeks post-procedure)
  Number of Serious Adverse Events (SAEs) associated with bleeding related to the investigational device and/or radiofrequency ablation (RFA) procedure.
Severity of Bleeding-Related Adverse Events as Assessed by the Nashville Bleeding Scale | From Day 0 (Diagnostic Bronchoscopy and RFA Procedure) through End of Study (6-7 weeks post-procedure)
  Safety assessments for bleeding Adverse Events (AEs) related to the investigational device and/or radiofrequency ablation (RFA) procedure, graded using the Nashville bleeding scale.

SECONDARY OUTCOMES:
Total Number of Serious Adverse Events Related to the Investigational Device and/or RFA Procedure | From Day 0 (Diagnostic Bronchoscopy and RFA Procedure) through End of Study (6-7 weeks post-procedure)
  Total number of Serious Adverse Events (SAEs) related to the investigational device and/or radiofrequency ablation (RFA) procedure.
Total Number of Adverse Events Related to the Investigational Device and/or RFA Procedure | From Day 0 (Diagnostic Bronchoscopy and RFA Procedure) through End of Study (6-7 weeks post-procedure)
  Total number of Adverse Events (AEs) related to the investigational device and/or radiofrequency ablation (RFA) procedure.
Macroscopic and Microscopic Evidence of Ablation in the Resected Specimen | At Surgical Resection (7-14 Days Post-Procedure)
  Macroscopic and microscopic evidence of ablation in the resected specimen, assessed using standard histopathological methods (hematoxylin and eosin staining).
Percentage of Tumor Necrosis Within the Ablation Zone | At Surgical Resection (7-14 Days Post-Procedure)
  Visual estimation of histopathologic ablation completeness, defined as the percentage of tumor necrosis within the ablation zone, as determined by routine pathology reporting.
Histopathologic Complete Response (Absence of Viable Tumor Cells) Within the Ablation Zone | At Surgical Resection (7-14 Days Post-Procedure)
  Evaluation of macroscopic and microscopic necrosis within the ablation zone, defined as the absence of viable tumor cells within the ablated area (histopathologic complete response, hpCR), if reported as part of routine histological assessment. If applicable, the extent of necrosis into surrounding parenchyma or margin tissue will be noted.
Composite Descriptive Intra-Procedural Metrics During Bronchoscopic Cryo-assisted RFA | Day 0 (Diagnostic Bronchoscopy and RFA Procedure)
  Descriptive intra-procedural metrics collected during the bronchoscopic cryo-assisted radiofrequency ablation (RFA) procedure, including total ablation time (minutes), number of cryoRFA activations (energy applications), electrical parameters of energy delivered (if available), number of probe repositionings within the lesion, and estimated ablation zone size (millimeters) derived from intraoperative imaging when obtained as part of routine clinical practice. These measures are collected for descriptive characterization of procedural performance and are not intended for separate outcome analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Raemistrasse, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to local data protection requirements.

REFERENCES:
- [Background] Signoretti M, Valente R, Repici A et al. Endoscopy-guided ablation of pancreatic lesions: Technical possibilities and clinical outlook. World J Gastrointest Endosc 2017; 9: 41-54
- [Background] Dabizzi E, Testoni SG, Barbera M et al. 484 EUS-GUIDED CRYOTHERM ABLATION OF STAGE III PANCREATIC ADENOCARCINOMA: A PRELIMINARY RADIOLOGICAL PERSPECTIVE. Gastrointest Endosc 2018; 87: AB84
- [Background] Testoni SGG, Petrone MC, Reni M et al. EUS-guided ablation with the HybridTherm Probe as second-line treatment in patients with locally advanced pancreatic ductal adenocarcinoma: A case-control study. Endosc Ultrasound 2022; 11: 383-392
- [Background] Testoni SGG, Petrone MC, Reni M et al. Efficacy of Endoscopic Ultrasound-Guided Ablation with the HybridTherm Probe in Locally Advanced or Borderline Resectable Pancreatic Cancer: A Phase II Randomized Controlled Trial. Cancers (Basel) 2021; 13
- [Background] Arcidiacono PG, Carrara S, Reni M et al. Feasibility and safety of EUS-guided cryothermal ablation in patients with locally advanced pancreatic cancer. Gastrointest Endosc 2012; 76: 1142-1151
- [Background] Ahmed M, Liu Z, Afzal KS et al. Radiofrequency ablation: effect of surrounding tissue composition on coagulation necrosis in a canine tumor model. Radiology 2004; 230: 761-767
- [Background] International Conference on Harmonization (ICH) Guideline for Good Clinical Practice E6(R2), (www.ich.org).
- [Background] Strahlenschutzverordnung (StSV) vom 26. April 2017 / Ordonnance sur la radioprotection (ORaP) du 26 avril 2017 / Ordinanza sulla radioprotezione (ORaP) del 26 aprile 2017
- [Background] WHO, International Clinical Trials Registry Platform (ICTRP) (http://www.who.int/ictrp/en/)
- [Background] EN ISO 14971: Application of risk management to medical devices (www.iso.org)
- [Background] EN ISO 10993: Biological evaluation of medical devices (www.iso.org)
- [Background] EN ISO 14155: Clinical investigation of medical devices for human subjects - Good clinical practice (www.iso.org)
- [Background] MDCG 2020-10/1 Safety reporting in clinical investigations of medical devices under the Regulation (EU) 2017/745 (https://ec.europa.eu/health/sites/health/files/md_sector/docs/md_mdcg_2020-10-1_guidance_safety_reporting_en.pdf)
- [Background] MDCG 2024-3 Guidance on content of the Clinical Investigation Plan for clinical investigations of medical devices
- [Background] Medical Device Regulation (EU) 2017/745 of 5 April 2017 (MDR)
- [Background] Medizinprodukteverordnung (MepV) vom 17. Oktober 2001 / Ordonnance sur les dispositifs médicaux (ODim) du 17 octobre 2001 / Ordinanza relativa ai dispositivi medici (ODmed) del 17 ottobre 2001
- [Background] Verordnung über klinische Versuche mit Ausnahme klinischer Versuche mit Medizinprodukten (Verordnung über klinische Versuche, KlinV) vom 20. September 2013 / Ordonnance sur les essais cliniques hors essais cliniques de dispositifs médicaux (Ordonnance sur les essais cliniques, OClin) du 20 septembre 2013. Ordinanza sulle sperimentazioni cliniche ad eccezione delle sperimentazioni cliniche con dispositivi medici (Ordinanza sulle sperimentazioni cliniche, OSRUm) del 20 settembre 2013
- [Background] Verordnung über klinische Versuche mit Medizinprodukten (KlinV-Mep) vom 1. Juli 2020 / Ordonnance sur les essais cliniques de dispositifs médicaux (OClin-Dim) du 1er juillet 2020 /. Ordinanza sulle sperimentazioni cliniche con dispositivi medici (OSRUm-Dmed) del 1 luglio 2020
- [Background] Humanforschungsgesetz, HFG Bundesgesetz über die Forschung am Menschen (Bundesgesetz über die Forschung am Menschen, HFG) vom 30. September 2011/ Loi fédérale relative à la recherche sur l'être humain (loi relative à la recherche sur l'être humain, LRH) du 30 septembre 2011 / Legge federale concernente la ricerca sull'essere umano (Legge sulla ricerca umana, LRUm) del 30 settembre 2011
- [Background] Steinfort DP, Herth FJF. Bronchoscopic treatments for early-stage peripheral lung cancer: Are we ready for prime time? Respirology 2020; 25: 944-952
- [Background] Koizumi T, Tsushima K, Tanabe T et al. Bronchoscopy-Guided Cooled Radiofrequency Ablation as a Novel Intervention Therapy for Peripheral Lung Cancer. Respiration 2015; 90: 47-55
- [Background] Tanabe T, Koizumi T, Tsushima K et al. Comparative registry of three different catheters for CT imaging-bronchoscopy-guided radiofrequency ablation as a potential and novel interventional therapy for lung cancer. Chest 2010; 137: 890-897
- [Background] Ishiwata T, Motooka Y, Ujiie H et al. Endobronchial ultrasound-guided bipolar radiofrequency ablation for lung cancer: A first-in-human clinical trial. The Journal of Thoracic and Cardiovascular Surgery 2022
- [Background] Koizumi T, Kobayashi T, Tanabe T et al. Clinical experience of bronchoscopy-guided radiofrequency ablation for peripheral-type lung cancer. Case Rep Oncol Med 2013; 2013: 515160
- [Background] Steinfort DP, Antippa P, Rangamuwa K et al. Safety and Feasibility of a Novel Externally Cooled Bronchoscopic Radiofrequency Ablation Catheter for Ablation of Peripheral Lung Tumours: A First-In-Human Dose Escalation Registry. Respiration 2023; 102: 211-219
- [Background] Xie F, Zheng X, Xiao B et al. Navigation Bronchoscopy-Guided Radiofrequency Ablation for Nonsurgical Peripheral Pulmonary Tumors. Respiration 2017; 94: 293-298
- [Background] Steinke K, King J, Glenn D et al. Pulmonary hemorrhage during percutaneous radiofrequency ablation: a more frequent complication than assumed? Interact Cardiovasc Thorac Surg 2003; 2: 462-465
- [Background] Vaughn C, Mychaskiw G, Sewell P. Massive hemorrhage during radiofrequency ablation of a pulmonary neoplasm. Anesth Analg 2002; 94: 1149-51; table of contents
- [Background] Vogl TJ, Eckert R, Naguib NNN et al. Thermal Ablation of Colorectal Lung Metastases: Retrospective Comparison Among Laser-Induced Thermotherapy, Radiofrequency Ablation, and Microwave Ablation. AJR Am J Roentgenol 2016; 207: 1340-1349
- [Background] Aufranc V, Farouil G, Abdel-Rehim M et al. Percutaneous thermal ablation of primary and secondary lung tumors: Comparison between microwave and radiofrequency ablation. Diagn Interv Imaging 2019; 100: 781-791
- [Background] Grasso RF, Bernetti C, Pacella G et al. A comparative analysis of thermal ablation techniques in the treatment of primary and secondary lung tumors: a single-center experience. Radiol Med 2022; 127: 714-724
- [Background] Shi F, Li G, Zhou Z et al. Microwave ablation versus radiofrequency ablation for the treatment of pulmonary tumors. Oncotarget 2017; 8: 109791-109798
- [Background] Chi J, Ding M, Shi Y et al. Comparison registry of computed tomography-guided radiofrequency and microwave ablation for pulmonary tumors: A retrospective, case-controlled observational registry. Thorac Cancer 2018; 9: 1241-1248
- [Background] Iezzi R, Larici AR, Posa A et al. Percutaneous radiofrequency ablation using internally cooled wet electrodes for the treatment of patients with lung tumors. Eur Rev Med Pharmacol Sci 2019; 23: 6554-6561
- [Background] Mu L, Pan T, Lyu N et al. CT-guided percutaneous radiofrequency ablation for lung neoplasms adjacent to the pericardium. Lung Cancer 2018; 122: 25-31
- [Background] Yang Q, Luo LC, Li FM et al. Survival outcomes of radiofrequency ablation compared with surgery in patients with early-stage primary non-small-cell lung cancer: A meta-analysis. Respir Investig 2022; 60: 337-344
- [Background] Rempp H, Voigtlander M, Clasen S et al. Increased ablation zones using a cryo-based internally cooled bipolar RF applicator in ex vivo bovine liver. Invest Radiol 2009; 44: 763-768
- [Background] Baere T de, Tselikas L, Catena V et al. Percutaneous thermal ablation of primary lung cancer. Diagn Interv Imaging 2016; 97: 1019-1024
- [Background] Lencioni R, Crocetti L, Cioni R et al. Response to radiofrequency ablation of pulmonary tumours: a prospective, intention-to-treat, multicentre clinical trial (the RAPTURE registry). Lancet Oncol 2008; 9: 621-628
- [Background] Dupuy DE, Zagoria RJ, Akerley W et al. Percutaneous radiofrequency ablation of malignancies in the lung. AJR Am J Roentgenol 2000; 174: 57-59
- [Background] Callister MEJ, Baldwin DR, Akram AR et al. British Thoracic Society guidelines for the investigation and management of pulmonary nodules. Thorax 2015; 70 Suppl 2: ii1-ii54
- [Background] Postmus PE, Kerr KM, Oudkerk M et al. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol 2017; 28: iv1-iv21
- [Background] Langer T. Prävention, Diagnostik, Therapie und Nachsorge des Lungenkarzinoms 2022
- [Background] Al-Alem I, Pillai K, Akhter J et al. Heat sink phenomenon of bipolar and monopolar radiofrequency ablation observed using polypropylene tubes for vessel simulation. Surg Innov 2014; 21: 269-276
- [Background] Liu Z, Ahmed M, Weinstein Y et al. Characterization of the RF ablation-induced 'oven effect': the importance of background tissue thermal conductivity on tissue heating. Int J Hyperthermia 2006; 22: 327-342
- [Background] Palussière J, Catena V, Buy X. Percutaneous thermal ablation of lung tumors - Radiofrequency, microwave and cryotherapy: Where are we going? Diagn Interv Imaging 2017
- [Background] Hinshaw JL, Lubner MG, Ziemlewicz TJ et al. Percutaneous tumor ablation tools: microwave, radiofrequency, or cryoablation--what should you use and why? Radiographics 2014; 34: 1344-1362
- [Background] Dupuy DE, Zuromski J, Pennathur A. Ablation for treating small pulmonary nodules: radiologic and surgical approach and perspectives. Curr Chall Thorac Surg 2022; 4: 40
- [Background] Long G, Bakos G, Shires PK et al. Histological and finite element analysis of cell death due to irreversible electroporation. Technol Cancer Res Treat 2014; 13: 561-569
- [Background] Megan E. Daly, Navneet Singh, Nofisat Ismaila et al. Management of Stage III Non-Small-Cell Lung Cancer: ASCO Guideline
- [Background] Howington JA, Blum MG, Chang AC et al. Treatment of stage I and II non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest 2013; 143: e278S-e313S
- [Background] American Cancer Society. Cancer Facts & Figures 2023; 2023
- [Background] Sung H, Ferlay J, Siegel RL et al. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin 2021; 71: 209-249
- [Background] Declaration of Helsinki, Version October 2013 (http://www.wma.net)